CLINICAL TRIAL: NCT00874302
Title: A Phase III, Open Label, Randomized, Multicenter Study Evaluating the Safety and Efficacy of 25 mg and 50 mg Doses of Proellex to Assess Recurrence of Symptoms in the Treatment of Symptomatic Uterine Fibroids
Brief Title: Safety and Efficacy of 25 and 50 mg Doses of Proellex® in Treating the Recurrence of Uterine Fibroid Symptoms
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated for safety and the FDA put the study on hold for safety.
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZPU-306
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Uterine Fibroids
Keywords: Uterine fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 25 mg (Experimental): 25 mg Proellex
  Interventions: Drug: Proellex
- 50 mg (Experimental): 50 mg Proellex
  Interventions: Drug: Proellex

INTERVENTIONS:
Drug: Proellex — One 25mg capsule taken orally once every day.
  Other Names: Telapristone acetate
  Arms: 25 mg
Drug: Proellex — Two 25mg capsules Proellex (50mg) taken orally once every day
  Other Names: Telapristone acetate
  Arms: 50 mg

SUMMARY:
Subjects with symptomatic uterine fibroids will be enrolled and will receive daily oral study medication for 4 months. This will be followed by a 6 month off-drug interval until there is a return of significant symptomatology. If they experience symptoms of a certain severity, the subject will enter a second 4 month treatment cycle and then a follow-up period.

DETAILED DESCRIPTION:
Subjects with documented symptomatic uterine fibroids will be enrolled in the study. Following screening, subjects will receive daily oral study medication and will be assessed monthly for a 4 month treatment cycle. This first cycle will be followed by an off-drug interval until there is a return of significant symptomatology. Subjects will be followed for up to six (6) months post-treatment. If their lack of symptoms does not qualify them for a second cycle of treatment, they will be discharged from the study. If they experience symptoms of a certain severity, the subject will enter a second 4 month treatment cycle and then a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* At least one uterine fibroid must be identifiable and measurable by Transvaginal Ultrasound (TVU)
* Subject must have uterine fibroid-associated symptoms during the-screening visit
* Subject has menstrual cycle lasting from 20 to 40 days
* Other inclusion criteria may apply

Exclusion Criteria:

* Post-menopausal women or women likely to become post-menopausal during the study
* Subject with a significant organ abnormality or disease (based on the Investigator's judgment) that would in the opinion of the Investigator exclude the subject from participating
* Subject with any medical condition that, in the opinion of the Investigator, is not compatible with study procedures or which would prevent the subject from starting or completing the study, or interfere with the subject participating in this study.
* Subject who has had an acute illness within five days of study medication administration
* Subject with endometrial thickness of ≥ 18 mm on screening ultrasound or historically
* Subject with an abnormal screening endometrial biopsy including the presence of Endometrial Intraepithelial Neoplasia (EIN)
* Subject with an abnormal DEXA scan with a diagnosis or indication of osteoporosis at screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of 25 and 50 mg Proellex administered once daily for two treatment cycles | Four months each cycle

SECONDARY OUTCOMES:
To evaluate the efficacy of two different doses of Proellex used for the treatment of symptomatic uterine fibroids | Two, 4 month cycles

CONTACTS AND LOCATIONS:
Overall Officials: Andre van As, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (20):
- United States (13):
  - Genesis Center for Clinical Research, San Diego, California
  - Physician Care Clinical Research, LLC, Sarasota, Florida
  - Atlanta Women's Research Inst., Atlanta, Georgia
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - York Clinical Consulting, Marrero, Louisiana
  - Female Pelvic Medicine, Grand Rapids, Michigan
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - Clinical Trials of America, Eugene, Oregon
  - Thomas Jefferson University - Jefferson Center for Women's Medical Specialties, Philadelphia, Pennsylvania
  - Women's Care Center, PLC Research Memphis Associates, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Willowbend Health & Wellness Associates, Plano, Texas
- Brazil (7):
  - Cepeme/Cerfahc, Curitiba, Paraná
  - Brazilmed, São Paulo, São Paulo
  - Universidade Federal de São Paulo - UNIFESP, São Paulo, São Paulo
  - Hospital dos Servidores Públicos de SP, São Paulo, São Paulo
  - Hospital Heliópolis, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
  - Vox Femina, Jundiaí